CLINICAL TRIAL: NCT04179162
Title: Phase I/II Trial of Bacillus Calmette-Guérin (BCG) and Intravesical Gemcitabine for Patients With BCG-Relapsing High-Grade Non-Muscle Invasive Bladder Cancer
Brief Title: Bacillus Calmette-Guérin (BCG) and Gemcitabine in People With High-Grade Non-Muscle Invasive Bladder Cancer That Came Back After BCG Treatment
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-374
Record Dates: First submitted 2019-11-25; First posted 2019-11-27 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Non-Muscle Invasive Bladder Cancer (NMIBC)
Keywords: Bacillus Calmette-Guérin (BCG); Gemcitabine; 19-374
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Intervention Model Description: This is a phase I/II trial of intravesical gemcitabine given between doses of BCG in patients who have relapsing but BCG-responsiveNon-Muscle Invasive Bladder Cancer (NMIBC).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bacillus Calmette-Guérin (BCG) and Gemcitabine (Experimental): Eligible patients will receive combination intravesical chemoimmunotherapy. Treatment is sequential, with twice-weekly intravesical gemcitabine given at weeks 1, 4, 7, and 10, for a total of 8 doses, administered in a standard fashion. In phase I, the dose of gemcitabine will depend on the dose level being assessed for the determination of the MTD. phase II, 1 dose level will be given (the MTD from phase I). Fixed doses of once-weekly intravesical BCG therapy (TICE strain, 50 mg) will be given at weeks 2 (+/- 2 days), 3 (+/- 2 days), 5 (+/- 2 days), 6 (+/- 2 days), 8 (+/- 2 days), and 9 (+/- 2 days), for a total of 6 doses, also administered in a standard fashion. All intravesical therapy will be administered in the chemotherapy suite on an outpatient basis, in accordance with standard clinical practice. Intravesical therapies will be retained in the bladder for up to 2 h (BCG) or 1 h (gemcitabine), or as tolerated.
  Interventions: Drug: Bacillus Calmette-Guérin (BCG); Drug: Gemcitabine

INTERVENTIONS:
Drug: Bacillus Calmette-Guérin (BCG) — Patients will receive once-weekly intravesical BCG therapy (TICE strain, 50 mg) at weeks 2 (+/- 2 days), 3 (+/- 2 days), 5 (+/- 2 days), 6(+/- 2 days), 8 (+/- 2 days), and 9 (+/- 2 days).
Drug: Gemcitabine — Patients will receive gemcitabine at their specified dose level, given in a twice weekly fashion, with 72 to 96 h (+/- 1 day) between doses, at weeks 1, 4, 7, and 10.

SUMMARY:
This study will test the safety of BCG and gemcitabine in people who have BCG-relapsing Non-Muscle Invasive Bladder Cancer (NMIBC). The researchers will test increasing doses of gemcitabine to find the highest dose that causes few or mild side effects when combined with BCG. The study will also look at whether this combination of drugs is effective in treating BCG-relapsing NMIBC.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent for persistent high-grade NMIBC Ta/T1/Tis (Ta/T1 with CIS is preferred, but not required) within 24 months of the last treatment with BCG (with or without IFN)

  o Up to 26 months from the last BCG treatment is allowed for the treating physician to perform a transurethral resection of bladder tumor (TURBT) so long as there is evidence of recurrent disease (by positive cytology, imaging, or office cystoscopy) within 24 months of last BCG transurethral resection of bladder tumor (TURBT)
* Pathologic confirmation of stage, grade, and urothelial histology by the Department of Pathology at MSK
* All visible papillary lesions macroscopically resected within 60 days of treatment initiation
* Absence of urothelial carcinoma involving the upper urinary tract (documented by radiological imaging or ureteroscopy) within 12 months from the start of treatment
* Receipt of restaging transurethral resection (TUR) for any tumor with invasion into the lamina propria (HGT1) as part of standard care
* Age ≥18 years
* Karnofsky performance status ≥60%
* Informed consent

Exclusion Criteria:

* Positive pregnancy test
* Known contraindications to BCG

  * History of systemic hypersensitivity reaction or history of febrile systemic BCG reaction
  * Febrile illness or persistent gross hematuria
  * Active tuberculosis
  * Immunosuppression due to congenital or acquired immune deficiency, concurrent immune suppressive disease, systemic cancer therapy, or chronic immunosuppressive therapy other than topical or inhaled corticosteroids
* History of or currently being treated for muscle-invasive (i.e., stage T2 or higher) or metastatic urothelial cell carcinoma
* Evidence of concurrent extravesical (i.e., urethra, ureter, or renal pelvis) urothelial cell carcinoma
* BCG-unresponsive NMIBC as defined by the FDA:

  * HGT1 within 3 months after an induction BCG course (received ≥5 of 6 doses)
  * Persistent or recurrent high-grade NMIBC (Tis, Ta, T1) within 6 months of ≥5 of 6 doses of induction BCG therapy and ≥2 of 3 doses of maintenance BCG therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
evaluate the MTD (Phase I) | 1 year
  Describe the toxicities by frequency and by grade.This study will use CTCAE version 5.0 for toxicity and serious adverse event reporting.
proportion of patients who are disease free | 6 months after the start of treatment
  Will be assessed by both urine cytology and cystoscopy at 6 months after initiation of therapy. Disease free (i.e., complete treatment response) is defined as no evidence of disease (negative cytology and cystoscopy).

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Pietzak, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Hartford Healthcare (Data Collection), Hartford, Connecticut
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm